CLINICAL TRIAL: NCT03311373
Title: A Randomized, Open-label, Single-dose, Single-center, Crossover Study in Healthy Subjects to Assess the Relative Bioavailability of PT010 Administered With and Without a Spacer, and With and Without Oral Charcoal
Brief Title: A Randomized, Open-label, Single-dose, Single-center, Crossover Study in Healthy Subjects to Assess the Relative Bioavailability of PT010
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PT010011
Record Dates: First submitted 2017-10-11; First posted 2017-10-17 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — OOS-A regimen; Regimen B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Period 1 (Experimental): Test Formulation (Regimen B or D) or Reference Formulation (Regimen A or C)
  Interventions: Drug: Regimen A; Drug: Regimen B; Drug: Regimen C; Drug: Regimen D
- Treatment Period 2 (Experimental): Test Formulation (Regimen (B or D) or Reference Formulation (Regimen A or C)
  Interventions: Drug: Regimen A; Drug: Regimen B; Drug: Regimen C; Drug: Regimen D
- Treatment Period 3 (Experimental): Test Formulation (Regimen (B or D) or Reference Formulation (Regimen A or C)
  Interventions: Drug: Regimen A; Drug: Regimen B; Drug: Regimen C; Drug: Regimen D
- Treatment Period 4 (Experimental): Test Formulation (Regimen (B or D) or Reference Formulation (Regimen A or C)
  Interventions: Drug: Regimen A; Drug: Regimen B; Drug: Regimen C; Drug: Regimen D

INTERVENTIONS:
Drug: Regimen A — 2 inhalations BGF MDI; no spacer device; no oral charcoal - reference formulation/total systemic exposure
Drug: Regimen B — 2 inhalations BGF MDI; AeroChamber Plus Flow-Vu spacer device; no oral charcoal - test formulation/total systemic exposure
Drug: Regimen C — 2 inhalations BGF MDI; no spacer device; with oral charcoal - reference formulation/lung exposure
Drug: Regimen D — 2 inhalations BGF MDI; AeroChamber Plus Flow-Vu spacer device; with oral charcoal - test formulation/lung exposure

SUMMARY:
Randomized, Open-label, Single-dose, Single-center, Crossover Study in Healthy Subjects to Assess the Relative Bioavailability of PT010

DETAILED DESCRIPTION:
A Randomized, Open-label, Single-dose, Single-center, Crossover Study in Healthy Subjects to Assess the Relative Bioavailability of PT010 Administered With and Without a Spacer, and With and Without Oral Charcoal

ELIGIBILITY:
Key Inclusion Criteria:

* Signed and dated Independent Ethics Committee (IEC)/Institutional Review Board (IRB)-approved Informed Consent Form (ICF) before any protocol-specific screening procedures are performed
* Male and female subjects 18 to 40 years of age, inclusive
* Be in good general health as determined by a thorough medical history and physical examination, ECG, vital signs, and clinical laboratory evaluation
* Non-childbearing potential (ie, physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal, or surgically sterile
* Male subjects who are sexually active must agree to use a double-barrier method of contraception (condom with spermicide) from the first dose of randomized study drug until 2 weeks after their last dose, and must not donate sperm during their study participation period
* Screening laboratory tests must be within normal range or determined to not be clinically significant by the Investigator.
* Demonstrate correct MDI administration technique

Key Exclusion Criteria:

* For female subjects, a positive serum human chorionic gonadotropin (hCG) test at screening or a positive urine hCG at admission for any of the 4 Treatment Periods
* Subjects with clinically significant neurologic, cardiovascular, hepatic, renal, endocrinologic, pulmonary, hematological, psychiatric, or other medical illness that would interfere with participation in this study
* Subjects who have cancer that has not been in complete remission for at least 5 years
* Male subjects with a trans-urethral resection of the prostate or full resection of the prostate within 6 months prior to screening
* Subjects with bladder neck obstruction or urinary retention that is clinically significant in the opinion of the Investigator
* History of substance-related disorders (with the exception of caffeine-related and nicotine-related disorders) within 1 year of screening
* History of smoking or the use of nicotine-containing products within 3 months of screening by self-reporting
* A positive alcohol breathalyzer or urine drug screen for drugs of abuse at screening or at the beginning of each Treatment Period
* Treatment with any prescription or non-prescription drugs including vitamins, herbal, and dietary supplements for 28 days or 5 half-lives, whichever is longer, before study drug use
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to the beginning of the screening Period
* Subjects with any flu-like syndrome or other respiratory infections within 2 weeks of drug administration or who have been vaccinated with an attenuated live virus within 4 weeks of drug administration
* Any other condition and/or situation that causes the Investigator to deem a subject unsuitable for the study (eg, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study-related procedures)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M. Dorinsky, MD, Study Director — Pearl Therapeutics, Inc.
Locations (1):
- Pearl Investigative Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Dorinsky P, DePetrillo P, DeAngelis K, Trivedi R, Darken P, Gillen M. Relative Bioavailability of Budesonide/Glycopyrrolate/Formoterol Fumarate Metered Dose Inhaler Administered With and Without a Spacer: Results of a Phase I, Randomized, Crossover Trial in Healthy Adults. Clin Ther. 2020 Apr;42(4):634-648. doi: 10.1016/j.clinthera.2020.02.012. Epub 2020 Apr 3. PMID 32253054
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=PT010011&attachmentIdentifier=101b3e8b-ad61-40b9-a1b0-4edfb4c6fb48&fileName=PT010011_SAP__v1.0_16J_Jan_2018_Redacted_Final_PDF-A.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=PT010011&attachmentIdentifier=9d004324-7532-460f-8551-bfd83a9ea40d&fileName=PT010011_Protocol_v1.0_11Sep2017__Redacted_Final-PDF-A.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States from November 2017 to December 2017.
Pre-assignment Details: Elig subj. received single dose of BGF MDI (Budesonide, Glycopyrronium, and Formoterol Fumarate metered dose inhaler) 320/28.8/9.6 μg as:
  Regimen A: BGF MDI w/out spacer, w/out charcoal Regimen B: BGF MDI with spacer, w/out charcoal Regimen C: BGF MDI w/out spacer, with charcoal Regimen D: BGF MDI with spacer, with charcoal
Groups:
- All Regimens: BGF MDI 320/28.8/9.6 μg
Period: Overall Study
Arm/Group | All Regimens
Started | 56
Completed | 47
Not Completed | 9
Not completed — Adverse Event | 1
Not completed — Protocol Discontinuation Criteria | 3
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.9 (5.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 34
  Female | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 47
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)-Budesonide
Description: Maximum plasma concentration (Cmax) per Regimen
Time Frame: Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 12 and 24 h post-dose
Population: PK Population: All subjects in the Safety Population for whom at least one of the primary PK parameters for a given analyte could be calculated and who had no important protocol deviations thought to impact the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- Regimen B: BGF MDI 320/28.8/9.6 μg with a spacer device and without charcoal
- Regimen A: BGF MDI 320/28.8/9.6 μg without spacer device and without charcoal
- Regimen C: BGF MDI 320/28.8/9.6 μg without a spacer device and with charcoal
- Regimen D: BGF MDI 320/28.8/9.6 μg with a spacer device and with charcoal
Arm/Group | Regimen B | Regimen A | Regimen C | Regimen D
Number analyzed (Participants) | 52 | 52 | 52 | 52
pg/mL | 702.3 (46.4) | 452.6 (74.6) | 340.0 (117.1) | 612.0 (74.0)

2. Primary Outcome: Maximum Plasma Concentration (Cmax)-Glycopyrronium
Description: Maximum plasma concentration (Cmax) per Regimen
Time Frame: Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Regimen B | Regimen A | Regimen C | Regimen D
Number analyzed (Participants) | 52 | 52 | 51 | 51
pg/mL | 47.7 (73.3) | 19.0 (131.0) | 17.1 (181.7) | 42.1 (65.4)

3. Primary Outcome: Maximum Plasma Concentration (Cmax)-Formoterol
Description: Maximum plasma concentration (Cmax) per Regimen
Time Frame: Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Regimen B | Regimen A | Regimen C | Regimen D
Number analyzed (Participants) | 52 | 52 | 51 | 51
pg/mL | 18.1 (58.4) | 10.8 (66.3) | 8.3 (98.6) | 17.9 (48.1)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 the Time of the Last Measurable Plasma Concentration (AUC0-tlast)-Budesonide
Description: Each treatment period is equal to assigned regimen
Time Frame: Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Regimen B | Regimen A | Regimen C | Regimen D
Number analyzed (Participants) | 52 | 52 | 52 | 52
h*pg/mL | 1934.0 (54.9) | 1452.8 (66.0) | 823.9 (121.2) | 1618.5 (74.9)

5. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 the Time of the Last Measurable Plasma Concentration (AUC0-tlast)-Glycopyrronium
Description: Each treatment period is equal to assigned regimen
Time Frame: Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Regimen B | Regimen A | Regimen C | Regimen D
Number analyzed (Participants) | 52 | 52 | 51 | 51
h*pg/mL | 74.3 (96.4) | 48.1 (122.4) | 19.8 (325.0) | 69.2 (85.2)

6. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 the Time of the Last Measurable Plasma Concentration (AUC0-tlast)-Formoterol
Description: Each treatment period is equal to assigned regimen
Time Frame: Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Regimen B | Regimen A | Regimen C | Regimen D
Number analyzed (Participants) | 52 | 52 | 51 | 51
h*pg/mL | 35.9 (97.5) | 37.0 (88.7) | 8.9 (471.8) | 33.1 (71.3)

7. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)-Budesonide
Description: Each treatment period is equal to assigned regimen
Time Frame: Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h (hour)
Arm/Group | Regimen B | Regimen A | Regimen C | Regimen D
Number analyzed (Participants) | 52 | 52 | 52 | 52
h (hour) | 0.33 [0.10 to 1.00] | 0.33 [0.10 to 2.00] | 0.33 [0.10 to 2.00] | 0.33 [0.10 to 1.00]

8. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)-Glycopyrronium
Description: Each treatment period is equal to assigned regimen
Time Frame: Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h (hour)
Arm/Group | Regimen B | Regimen A | Regimen C | Regimen D
Number analyzed (Participants) | 52 | 52 | 51 | 51
h (hour) | 0.03 [0.03 to 0.67] | 0.03 [0.03 to 4.00] | 0.03 [0.03 to 0.67] | 0.03 [0.03 to 0.10]

9. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)-Formoterol
Description: Each treatment period is equal to assigned regimen
Time Frame: Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h (hour)
Arm/Group | Regimen B | Regimen A | Regimen C | Regimen D
Number analyzed (Participants) | 52 | 52 | 51 | 51
h (hour) | 0.10 [0.03 to 0.67] | 0.10 [0.03 to 4.00] | 0.10 [0.03 to 0.67] | 0.10 [0.03 to 0.33]

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 Extrapolated to Infinity (AUC0-∞);-Budesonide
Description: Each treatment period is equal to assigned regimen
Time Frame: Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Regimen B | Regimen A | Regimen C | Regimen D
Number analyzed (Participants) | 49 | 51 | 49 | 48
h*pg/mL | 2132.1 (40.9) | 1491.8 (64.4) | 823.9 (121.2) | 1806.2 (39.1)

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 Extrapolated to Infinity (AUC0-∞);-Glycopyrronium
Description: Each treatment period is equal to assigned regimen
Time Frame: Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Regimen B | Regimen A | Regimen C | Regimen D
Number analyzed (Participants) | 5 | 4 | 7 | 7
h*pg/mL | 40.4 (49.6) | 65.9 (44.7) | 15.2 (54.5) | 39.2 (96.5)

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 Extrapolated to Infinity (AUC0-∞);-Formoterol
Description: Each treatment period is equal to assigned regimen
Time Frame: 24 hrs
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Regimen B | Regimen A | Regimen C | Regimen D
Number analyzed (Participants) | 20 | 18 | 11 | 4
h*pg/mL | 63.2 (37.1) | 62.7 (62.2) | 62.6 (55.0) | 62.0 (42.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of administration of the first dose of study drug to the time of the follow-up telephone call, study termination, or study exit up to a total of approximately 12 weeks.
Description: Serious Adverse Events were collected from the time the subject signed informed consent throughout the treatment period and up to approximately 13 weeks, which includes screening and follow up (5-7 day period after study drug).
Arm/Group | Regimen B | Regimen A | Regimen C | Regimen D
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/52 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52 | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 4/53 | 1/52 | 4/52 | 4/52
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen B (N=53) | Regimen A (N=52) | Regimen C (N=52) | Regimen D (N=52)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT03311373/SAP_000.pdf
  • Study Protocol (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT03311373/Prot_001.pdf